CLINICAL TRIAL: NCT05440253
Title: Effectiveness of Dry Needling VS Ischaemic Compression on Latent Myofascial Myofascial Trigger Points in the Gluteus Medius in Patients With Patients With Non-specific Low Back Pain: a Randomised Clinical Trial
Brief Title: Effectiveness of Manual Therapy in Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 230622
Record Dates: First submitted 2022-06-23; First posted 2022-06-30 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Physiotherapy Specialty; Low Back Pain
Keywords: dry needling; low back pain; physiotherapy specialty; pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Dry Needling; Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dry needling group (Experimental)
  Interventions: Device: dry needling
- ischaemic compression group (Active Comparator)
  Interventions: Procedure: ischemic compression

INTERVENTIONS:
Device: dry needling — Dry needling of the trigger point of the gluteus medius in patients diagnosed with non-specific low back pain.
  Arms: dry needling group
Procedure: ischemic compression — Ischaemic trigger point compression of the gluteus medius in patients diagnosed with non-specific low back pain.
  Arms: ischaemic compression group

SUMMARY:
Low back pain affects many people and involves high medical costs. For this reason, we wish to test the efficacy of dry needling VS ischaemic compression in patients with non-specific low back pain. To this end, an investigation was carried out on 40 patients diagnosed with this ailment, divided into two groups by randomisation to assess the intensity of pain, range of movement, pain threshold to pressure and quality of life, measuring these variables prior to the intervention, immediately, at 48 hours and one week after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Presence of non-specific low back pain for more than six weeks.
* Presence of a palpable tight band nodule in the gluteus medius muscle.
* Presence of a hypersensitive or hyperirritable point in the tight band.
* Patients reporting local or referred pain in the area of the latent MGP after mechanical stimulation mechanical stimulation.

Exclusion Criteria:

* Surgeries in the lumbopelvic region.
* Diagnosis of herniated discs in the lumbar region.
* Positive cognitive screening according to the Pfeiffer questionnaire.
* Heterometrics.
* Age outside the range of 18 to 75 years.
* Ingested or injected anticoagulant or antiplatelet drugs.
* Systemic or local infection in the lumbar region.
* Pregnancy.
* Presence of fear of needles (belonephobia).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Pain | 1 week
  Visual Scale Analogue (0 minimum, 10 maximum).

SECONDARY OUTCOMES:
movement | 1 week
  Schober test (0 minimum, 45 maximun).
quality of life | 1 week
  Oswestry low back pain disability scale (0 minimum, 100% maximum; Between 0-20% minimal limitation or disability, 21-40% moderate limitation or disability, 41- 60% severe limitation or disability, 61-80% disabled and above 81% limitation or disability.
  60% severe limitation or disability, 61-80% disabled and above 81% maximum functional limitation or disability, 61-80% disabled and above 81% maximum functional limitation or disability.
  maximum functional limitation).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martinez de la Iglesia J, Duenas Herrero R, Onis Vilches MC, Aguado Taberne C, Albert Colomer C, Luque Luque R. [Spanish language adaptation and validation of the Pfeiffer's questionnaire (SPMSQ) to detect cognitive deterioration in people over 65 years of age]. Med Clin (Barc). 2001 Jun 30;117(4):129-34. doi: 10.1016/s0025-7753(01)72040-4. Spanish. PMID 11472684
- [Background] Kim HS, Lee JH, Kim IK. Intracellular glutathione level modulates the induction of apoptosis by delta 12-prostaglandin J2. Prostaglandins. 1996 Jun;51(6):413-25. doi: 10.1016/0090-6980(96)00047-0. PMID 8873236
- [Result] Perez-Palomares S, Jimenez-Sanchez C, Serrano-Herrero I, Herrero P, Calvo S. Is Instrumental Compression Equally Effective and Comfortable for Physiotherapists and Physiotherapy Students than Manual Compression? A Comparative Cross-Sectional Study. Int J Environ Res Public Health. 2021 Nov 18;18(22):12121. doi: 10.3390/ijerph182212121. PMID 34831877
- [Result] Aguilera FJ, Martin DP, Masanet RA, Botella AC, Soler LB, Morell FB. Immediate effect of ultrasound and ischemic compression techniques for the treatment of trapezius latent myofascial trigger points in healthy subjects: a randomized controlled study. J Manipulative Physiol Ther. 2009 Sep;32(7):515-20. doi: 10.1016/j.jmpt.2009.08.001. PMID 19748402
- [Result] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727
- [Result] Martin-Pintado-Zugasti A, Mayoral Del Moral O, Gerwin RD, Fernandez-Carnero J. Post-needling soreness after myofascial trigger point dry needling: Current status and future research. J Bodyw Mov Ther. 2018 Oct;22(4):941-946. doi: 10.1016/j.jbmt.2018.01.003. Epub 2018 Jan 17. PMID 30368339
- [Result] Martin-Pintado-Zugasti A, Rodriguez-Fernandez AL, Fernandez-Carnero J. Postneedling soreness after deep dry needling of a latent myofascial trigger point in the upper trapezius muscle: Characteristics, sex differences and associated factors. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):301-308. doi: 10.3233/BMR-150630. PMID 26406209
- [Result] Ziaeifar M, Arab AM, Karimi N, Nourbakhsh MR. The effect of dry needling on pain, pressure pain threshold and disability in patients with a myofascial trigger point in the upper trapezius muscle. J Bodyw Mov Ther. 2014 Apr;18(2):298-305. doi: 10.1016/j.jbmt.2013.11.004. Epub 2013 Nov 9. PMID 24725800